CLINICAL TRIAL: NCT04258904
Title: A Prospective Study of Dermatological Complications Associated With Continuous Subcutaneous Insulin Infusion and/or Continuous Glucose Monitoring in Pediatric Patients With Type 1 Diabetes
Brief Title: Prevention of Skin Problems With Diabetes Devices in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Jannet Svensson, MD, PhD, Assistant Professor, Copenhagen University Hospital at Herlev
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SkinProsp_29042019_v6
Record Dates: First submitted 2020-01-28; First posted 2020-02-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Type 1 Diabetes; Dermatologic Complication
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Skin Care Program
  Interventions: Combination Product: Skin Care Program
- Control (No Intervention): Usual Treatment

INTERVENTIONS:
Combination Product: Skin Care Program — The intervention consists of a Skin Care Program including neat information regarding dermatological complications to the device use, prevention of these and moisturizer to keep healthy skin.
  Arms: Intervention

SUMMARY:
A Cluster-controlled Intervention Trial regarding Prevention of Dermatological Complications towards use of Continuous glucose monitoring and insulin pumps in pediatric patients with Type 1 Diabetes. The patients will be followed prospectively with visits every 3rd month for the first year of initiation of device. Besides a standardized treatment plan if dermatological complications evolve, will be used.

DETAILED DESCRIPTION:
Background Unfortunately it has been shown earlier that dermatological complications are a huge challenge towards treatment with CSII and CGM in children. A preceding cross-sectional study in Danish patients showed that 90% of the 143 pediatric patients using CSII had experienced dermatological complications. Of those more than 60% currently had visible skin reaction due to the CSII. Dermatological complications to CSII were associated to atopic diseases and use of pump treatment for a longer period. For patients using CGM, 80% reported dermatological complications to the treatment, the most frequent being itching affecting more than 70%. Furthermore, 46% had at least one site with skin reaction due to CGM.

In the future, the use of artificial pancreas with closed-loop systems will still be dependent on the use of patches to fasten infu-sion sets and sensors. This skin complications poses a major challenge that must be investigated to reduce the overall burden of this chronic disease. The investigators have conducted a focus group study, which has given new insight into the perception of dermatological complications and further in-depth understanding of potential disease mechanisms regarding development of dermatological complications. No studies exist relating to prevention, consequences and treatment of dermatological complications in the setting of adhesive systems in T1D treatment.

Risk factors for development of dermatological complications are not well-known yet. Therefore, the investigators aim to create a possibly preventive screening tool based on a prospective study to guide future clinicians in whom patients are in risk of dermatological complications during use of CSII and CGM. This could help in guidance of which patients to give more information, preventive treatment or a more skin-sensitive CSII/CGM-system.

The hypothesis is that intensive information and proper skin care prior and during the initiation of CSII and CGM use, can reduce the dermatological

Study design This study is a prospective longitudinal study and will be the first longitudinal study concerning dermato-logical complications in a T1D population. It is a trial based on experience from pre-ceding cross-sectional study. The study is also a cluster-controlled intervention trial and will be the first interventional study regarding dermatological complications too. The intervention consists of intensive information about dermatological complications and possible preventive actions with skin moisturizing use. The cluster-controlling will include clusters defined by all patients from same de-partment. Patients enrolled from Herlev and Gentofte University Hospital will constitute the intervention group. Besides, a subgroup of the intervention group will be randomized to the ultrasound-skin-sites-intervention.

Justification for study design:

Dermatological complications construct a major challenge in diabetes technology especially among children and adolescents. To identify the modifiable or non-modifiable risk factors a prospective longitudinal study-design must be carried out. The longitudinal study-design will be combined with the interventional study to make the most of participants effort since the participants anyway will be investigated the first 12 months of their use of CSII and/or CGM/FGM. The interventional design could give important information regarding the possible effects of proper information and support regarding dermatological skin care and complications. And hopefully this could be a cheap way to reduce the dermatological complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 Diabetes
* Initiating either Insulin pump, Flash glucose monitorer or continuous glucose monitor

Exclusion Criteria:

*Language difficulties regarding Danish

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 236 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dermatological complications | Up to 12 months after inclusion
  Dermatological complications towards the devices will be assessed by clinical examination made by the investigator at visits every 3rd month and using a standardized scheme combined with self-reporting from the patients through diary forms if dermatological complications arise between visits. The incidence of dermatological complications through the time frame will be reported as primary outcome.

SECONDARY OUTCOMES:
Trans Epidermal Water Loss (TEWL): | Up to 12 months after inclusion
  TEWL value is a good measure of the leaky properties of the skin (the water evaporation rate). It is measured by Aquaflux AF2000 from Biox Systems

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Svensson, Principal Investigator — Department of Pediatrics, Herlev and Gentofte Hospital
Locations (1):
- Department of Pediatrics, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen FMW, Svensson J, Kinnander C, Berg AK. Ultrasound Detected Subcutaneous Changes in a Pediatric Cohort After Initiation of a New Insulin Pump or Glucose Sensor. Diabetes Technol Ther. 2023 Sep;25(9):622-630. doi: 10.1089/dia.2023.0137. Epub 2023 Jun 6. PMID 37279034